CLINICAL TRIAL: NCT01527058
Title: Radiation Dosimetry, Plasma Pharmacokinetics, Biodistribution, Safety and Diagnostic Performance of 68Ga-BNOTA-PRGD2 in Healthy Volunteers and Lung Cancer Patients
Brief Title: 68Ga-BNOTA-PRGD2 PET/CT in Healthy Volunteers and Lung Cancer Patients
Acronym: GRGDLC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM002
Record Dates: First submitted 2012-01-30; First posted 2012-02-06 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2014-11

CONDITIONS: Lung Cancer
Keywords: lung cancer; integrin receptor; 68Ga-BNOTA-PRGD2; PET/CT; efficacy and safety
MeSH Terms: conditions — Lung Neoplasms | interventions — 68gallium-BNOTA-PRGD2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-BNOTA-PRGD2 PET/CT scanning (Experimental): Determine if 68Ga-BNOTA-PRGD2 PET/CT is safe and effective method for imaging of lung cancer
  Interventions: Drug: 68Ga-BNOTA-PRGD2

INTERVENTIONS:
Drug: 68Ga-BNOTA-PRGD2 — Cancer patients, single intravenous bolus injection of nearly 111 MBq 68Ga-NOTA-PRGD2 on day one of the treatment period, dynamic whole-body PET/CT for determination of effective dose, kinetics of 68Ga-BNOTA-PRGD2 in blood, organs, and tumors
  Healthy volunteers, single intravenous bolus injection of nearly 111 MBq 68Ga-BNOTA-PRGD2 on day one of the treatment period, dynamic whole-body PET/CT for determination of effective dose, kinetics of 68Ga-BNOTA-PRGD2 in blood and organs
  Other Names: 68Ga-p-SCN-Bn-NOTA-PEG3-RGD2

SUMMARY:
This is an open-label dynamic whole-body PET/CT (positron emission tomography/computed tomography) study for investigation of radiation dosimetry, plasma pharmacokinetics, biodistribution, safety and diagnostic performance of 68Ga-BNOTA-PRGD2 in healthy volunteers and lung cancer patients. A single dose of nearly 111 MBq 68Ga-BNOTA-PRGD2 ( ≤ 40 µg BNOTA-PRGD2) will be intravenously injected into healthy volunteers and lung cancer patients. Visual and semiquantitative method will be used to assess the PET/CT images. Changes of blood pressure, pulse, respiration, temperature, routine blood and urine tests, serum alanine aminotransferase, albumin, and creatinine, and any adverse events will be collected from the volunteers. Adverse events will also be observed in the patients.

DETAILED DESCRIPTION:
Integrin αⅤβ3 is an important member of this receptor family and expressed preferentially on various types of tumor cells and the activated endothelial cells of tumor angiogenesis, but not or very low on the quiescent vessel cells and other normal cells. Therefore, the integrin αⅤβ3 receptor is becoming a valuable target for diagnosis and response evaluation of malignant tumors.

The tri-peptide sequence of arginine-glycine-aspartic acid (RGD) can specifically bind to the integrin αⅤβ3 receptor. Accordingly, a variety of radiolabeled RGD-based peptides have been developed for non-invasive imaging of integrin αⅤβ3 expression via positron emission tomography (PET) or single photon emission computed tomography (SPECT). Among all the RGD radiotracers studied, two PET imaging agents, 18F-Galacto-RGD and 18F-AH111585, have been investigated in clinical trials, and the results demonstrated that both radiotracers allowed the specific imaging of various types of tumors, and the tumor uptake correlated well with the expression of integrin αⅤβ3. Recently, series of RGD dimeric peptides with PEG linkers have been studied. The new types of RGD peptides showed much higher in vitro integrin αⅤβ3-binding affinity than the single RGD tri-peptide sequence, and importantly, they exhibited significantly increased tumor uptake and improved in vivo kinetics in animal models. As a representative, 68Ga-BNOTA-PRGD2 could be easily prepared and exhibited excellent in vivo behaviors in animal models. No adverse reactions are observed in animal models to date.

For the further interests in clinical translation of 68Ga-BNOTA-PRGD2, a open-label dynamic whole-body PET/CT study was designed to investigate radiation dosimetry, plasma pharmacokinetics, biodistribution, safety and diagnostic performance of 68Ga-BNOTA-PRGD2 in healthy volunteers and lung cancer patients. A single dose of nearly 111 MBq 68Ga-BNOTA-PRGD2 ( ≤ 40 µg BNOTA-PRGD2) will be intravenously injected into healthy volunteers and lung cancer patients. Visual and semiquantitative method will be used to assess the PET/CT images. Changes of blood pressure, pulse, respiration, temperature, routine blood and urine tests, serum alanine aminotransferase, albumin, and creatinine, and any adverse events will be collected from the volunteers. Adverse events will also be observed in the patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:

  * Males and females, ≥30 and ≤ 70 years old
* Cancer patients:

  * Males and females, ≥30 years old
  * CT and/or 18F-FDG PET/CT diagnosis in suspicion of primary or recurrent lung cancer.
  * The lung cancer will be histologically confirmed or results of histology will be available.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential
* Renal function: serum creatinine >3.0 mg/dL (270 μM/L)
* Liver function: any hepatic enzyme level more than 5 times upper limit of normal.
* Known severe allergy or hypersensitivity to IV radiographic contrast.
* Patients not able to enter the bore of the PET/CT scanner.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the Investigator, may significantly interfere with study compliance.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Visual and semiquantitative assessment of lesions and biodistribution | One year
  Visual analysis will be performed by consensus reading by at least 3 experienced nuclear medicine physician. The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake values (SUVs) of tumor and organs will be measured.

SECONDARY OUTCOMES:
Blood pressure | One year
  Blood pressure of healthy volunteers will be measured at three time points: right before injection, after scanning, and 24 hours after treatment.
Pulse | One year
  Pulse will be measured at three time points for each healthy volunteer: right before injection, after scanning, and 24 hours after treatment.
Respiration frequency | One year
  Respiration frequency will be measured at three time points for each healthy volunteer: right before injection, after scanning, and 24 hours after treatment.
Temperature | One year
  Temperature will be measured at three time points for each healthy volunteer: right before injection, after scanning, and 24 hours after treatment.
Routine blood test | One year
  Routine blood test of healthy volunteers will be measured at two time points: right before and 24 hours after treatment.
Routine urine test | One year
  Routine urine test of healthy volunteers will be measured at two time points: right before and 24 hours after treatment.
Serum alanine aminotransferase | One year
  Serum alanine aminotransferase of healthy volunteers will be measured at two time points: right before and 24 hours after treatment.
Serum albumin | One year
  Serum albumin of healthy volunteers will be measured at two time points: right before and 24 hours after treatment.
Serum creatinine | One year
  Serum creatinine of healthy volunteers will be measured at two time points: right before and 24 hours after treatment.
Adverse events collection | One year
  Adverse events within 5 days after the injection and scanning of healthy volunteers and patients will be followed and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, MD, Study Chair — Department of Nuclear Medicine, Peking Union Medical College Hospital, Chinese Academy of Medical Science
Locations (1):
- Department of Nuclear Medicine, Peking Union Medical College Hopital, Beijing, China

IPD SHARING:
Plan to Share IPD: No